CLINICAL TRIAL: NCT07153081
Title: Evaluating Wearable-supported Exercise Interventions for Reducing Postpartum Weight: a Randomized Controlled Trial
Brief Title: Wearable-Supported Exercise to Reduce Postpartum Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Bernard Chern Su Min, Head ＆ Senior Consultant, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIRB: Ref No.: 2017/3015
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Weight Change
Keywords: postpartum; physical activity; weight change; randomised controlled trial
MeSH Terms: conditions — Body Weight Changes; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized, single-center, unblinded intervention study with a 1:! allocation ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actigraphy watch intervention (Experimental): All the participants in the intervention group received an Actigraphy watch to wear all the time except for swimming and showering. Walking advises and motivational text messages will be sent to the study participants by the research team.
  Interventions: Device: Actigraphy watch intervention
- Standard care group (No Intervention): Walking advises and motivational text messages will be sent to the study participants by the research team.

INTERVENTIONS:
Device: Actigraphy watch intervention — Participants in this group only will be given an Actigraphy watch to track their physical activity levels.
  Arms: Actigraphy watch intervention

SUMMARY:
The aim of this study is to examine the effect of walking exercise in postpartum women and to evaluate the weight management intervention by using step tracker. The following hypotheses will be tested:

1. The intervention in postpartum women would reduce the retention of weight gained during pregnancy and lower the risk factors of chronic disease.
2. Step tracker is an effective tool in encouraging the postpartum women to do more physical activity.
3. Higher physical activity is recommended for postpartum women for healthy weight lost.

DETAILED DESCRIPTION:
Postpartum is an important phase in the reproductive years of women. Weight retention after childbirth can lead to chronic diseases (CD), including obesity, cardiovascular disease and other metabolic related diseases such as diabetes or high blood pressure. There are some studies suggesting that pedometer is useful to encourage women in increasing their physical activity.

We propose to evaluate the effects of physical activity intervention based on wearable steps tracker and optimal weight loss for postpartum women. It will be a pilot stratified randomized intervention study on 200 postpartum women at KK Women's and Children's Hospital. Women who are above 21 years old and had given birth between 6 weeks and 6 months before will be recruited under the study. Postpartum women who physically fit to participate in moderate intensity walking are eligible to participate in the study. Women who participated in other weight management or physical activity intervention projects will be excluded from the study. Study enrolment will be done at the Specialist Outpatient Clinics for postnatal check-ups.

This was 12-16 weeks randomized, single-center, unblinded intervention study (Figure 1). Participants were allocated in a 1:1 ratio to either the intervention group (Actigraphy watch) or the control group (no Actigraphy watch). All participants received the standard routine postpartum care, physical activity counselling with advice on walking and motivational messages. Randomization was done using sealed envelopes. Eligible participants had baseline measurements taken during the study enrolment and consent taking where anthropometric measurements, and blood samples were collected and various questionnaires were filled out to assess baseline demographics and lifestyle characteristics.

All the participants in the intervention group received an Actigraphy watch to wear all the time except for swimming and showering. Walking advises and motivational text messages will be sent to the study participants by the research team.

Data will be collected through questionnaires and clinical measurements. The questionnaires include socio-economic factors, and self-reported physical activity. Bio-physical measurements will be obtained from anthropometric measurements of participants, are collected from the participants at their follow-up time points. Objective physical activity will be collected using an Actigraphy watch.

ELIGIBILITY:
Inclusion Criteria:

1. Above 21 years old
2. Viable singleton pregnancies
3. Physically fit to participate in moderate intensity walking.
4. Term pregnancy without any sever pregnancy complications. -

Exclusion Criteria:

* 1. Blood-borne disease patients (e.g. HIV, hepatitis B & C) 2. Participated in other weight management or physical activity intervention projects.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women
Enrollment: 49 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
Weight change at the end of the intervention at 10 weeks postpartum | At 8-12 weeks postpartum from baseline (4-8 weeks postpartum)
  Using measured weight in kgs
Weight change at the end of the intervention at 14 weeks postpartum | At 12 to 16 weeks postpartum from baseline ( 4-8 weeks postpartum)
  Using measured weight in kgs

SECONDARY OUTCOMES:
Change in body mass index measures from baseline, 10 weeks postpartum and 14 weeks postpartum | Baseline (4-8 weeks postpartum), 10 weeks postpartum ( 8-12 weeks postpartum) and 14 weeks postpartum (12-16 weeks postpartum)
  Calculating body mass index (kg/m2) using height (m) and weight (kg) measures
Change in waist circumference measures from baseline, 10 weeks postpartum and 14 weeks postpartum | Baseline (4-8 weeks postpartum), 10 weeks (8-12 weeks postpartum) and 14 weeks (12-16 weeks postpartum)
  Using waist circumference measures in cm
Change in waist to hip ratio from baseline, 10 weeks and 14 weeks postpartum | Baseline 6 weeks postpartum (4-8 weeks postpartum), 10 weeks postpartum (8-12 weeks postpartum) and 14 weeks postpartum (12-16 weeks postpartum).
  Using waist circumference and hip measures
Change in body fat mass from baseline, 10 and 14 weeks postpartum | Baseline, 10 weeks postpartum (8-12 weeks postpartum) and 14 weeks (12-16 weeks postpartum)
  Using body fat mass percentage measured using the bioelectrical impedance analysis scale
Change in fasting lipid profile from baseline, 10 weeks and 14 weeks postpartum | Baseline, 10 weeks (8-12 week postpartum) and 14 weeks (12-16 weeks postpartum)
  Using fasting lipid profiles (total cholesterol, Low-density lipoprotein (LDL) cholesterol, High-density lipoprotein (HDL) cholesterol, triglycerides) of blood samples in mmol/L
Change in glucose homeostasis markers from baseline at 10 weeks and 14 weeks postpartum | Baseline, 10 weeks (8-12 weeks postpartum), and 14 weeks (12-16 weeks postpartum)
  Using fasting glucose and fasting insulin from blood samples in mmol/L
Change in blood pressure from baseline at 10 weeks and 14 weeks postpartum | At baseline, 10 weeks (8-12 weeks postpartum) and 14 weeks (12-16 weeks postpartum)
  Using measured systolic and diastolic blood pressure in mm/Hg
Change in self-reported frequency of moderate to vigorous physical activity at baseline, 10 weeks and 14 weeks | At baseline, 10 weeks (8-12 weeks postpartum) and 14 weeks (12-16 weeks postpartum).
  Self-reported data from the International Physical Activity Questionnaire (IPAQ) to assess frequency of moderate to vigorous physical activity.
Change in self-reported duration of moderate to vigorous physical activity at baseline, 10 weeks and 14 weeks | At baseline, 10 weeks (8-12 weeks postpartum) and 14 weeks (12-16 weeks postpartum).
  Self-reported data from the International Physical Activity Questionnaire (IPAQ) to assess duration of moderate to vigorous physical activity..
Change in duration of objective moderate to vigorous physical activity at baseline, 10 weeks and 14 weeks | Baseline, 10 weeks postpartum (8-12 weeks postpartum) and 14 weeks (12-16 weeks).
  MVPA will be assessed using an Actigraphy accelerometer Duration: Average daily/weekly minutes of MVPA (minutes per week).
Change in frequency of objective moderate to vigorous physical activity at baseline, 10 weeks and 14 weeks | Baseline, 10 weeks postpartum (8-12 weeks postpartum) and 14 weeks (12-16 weeks).
  MVPA will be assessed using an Actigraphy accelerometer Frequency: Number of days per week with ≥30 minutes of MVPA (days per week).

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Su Min Chern, MD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared due to privacy concerns and the potential risk of re-identification, especially in a small sample size or a highly specific population

REFERENCES:
- [Background] Maturi MS, Afshary P, Abedi P. Effect of physical activity intervention based on a pedometer on physical activity level and anthropometric measures after childbirth: a randomized controlled trial. BMC Pregnancy Childbirth. 2011 Dec 16;11:103. doi: 10.1186/1471-2393-11-103. PMID 22176722
- [Background] Davenport MH, Giroux I, Sopper MM, Mottola MF. Postpartum exercise regardless of intensity improves chronic disease risk factors. Med Sci Sports Exerc. 2011 Jun;43(6):951-8. doi: 10.1249/MSS.0b013e3182051155. PMID 21085038

DOCUMENTS (1):
  • Informed Consent Form (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT07153081/ICF_000.pdf